CLINICAL TRIAL: NCT01908998
Title: Influence of Supportive Sandals on Y-Balance Performance on Healthy Young Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Temple University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 21460
Record Dates: First submitted 2013-07-17; First posted 2013-07-26 (Estimated); Last update posted 2015-04-20 (Estimated); Status verified 2015-04

CONDITIONS: Y-balance Performance
Keywords: Y-Balance test
MeSH Terms: interventions — sandal wood oil-turmeric cream

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sandal (Active Comparator)
  Interventions: Other: Sandal

INTERVENTIONS:
Other: Sandal — Subjectes will be scored on the Y-Balance Test wearing an Orthaheel Sandal
  Other Names: Orthaheel Sandal

SUMMARY:
The Y-balance test is a lower extremity, dynamic test performed in single limb stance that measures a person's ability to reach in 3 directions. The test is typically conducted in barefoot. The purpose of this study is to assess the impact of footwear on Y-Balance test scores. The investigators hypothesize that by improving alignment and augmenting muscle mechanics, sandals with medial arch support may improve Y-Balance scores.

ELIGIBILITY:
Inclusion Criteria:

* Men or Women between the ages of 21 to 40 years, inclusive
* Grossly intact and symmetrical neuromuscular status
* Able to ambulate without difficult or pain
* Able to understand the information in the informed consent form
* willing and able to sign informed consent form

Exclusion Criteria:

* history of ankle sprain, Anterior cruciate ligament injury; recent hip, knee, foot or ankle pain within past 6 months
* Uncontrolled Heart (Hypertension; BP >= 140/90), Lung Disease (uncontrolled asthma or shortness of breath), or diabetes
* Nursing or pregnant
* Not willing or able to follow procedures specified by protocol and/or instructions of the study personnel
* Unable to fit into available shoe sizes

Ages: 21 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2013-07; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Y-Balance Test Score | Day 1
  Anterior, Posterior-medial and posterior-lateral maximum displacement (in cm) will be recorded as the best of three trials for each supportive limb in barefoot, supportive sandal and flip-flop

SECONDARY OUTCOMES:
Arch Height Index | Day 1
  An instrumented measure of arch height will be taken

OTHER OUTCOMES:
Malleolar Valgus Index | Day 1
  Malleolar valus testing will be performed to assess the structure of the hind foot
EMED-X | Day 1
  An EMED-X device will be used to assess plantar pressure when walking
GaitMatII | Day 1
  temporal and spatial foot fall parameters will be quantified with the GaitMatII.

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Pettineo, DPT, Principal Investigator — Temple University; Jinsup Song, DPM, Principal Investigator — Temple University
Locations (1):
- Temple University School of Podiatric Medicine, Philadelphia, Pennsylvania, United States